CLINICAL TRIAL: NCT04472767
Title: Phase 2 Study of Cabozantinib Combined With Ipilimumab/Nivolumab and Transarterial Chemoembolization (TACE) in Patients With Hepatocellular Carcinoma (HCC) Who Are Not Candidates for Curative Intent Treatment
Brief Title: Cabozantinib Combined With Ipilimumab/Nivolumab and TACE in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Farshid Dayyani, Associate Clinical Professor of Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20205807; UCI 19-49 (Other: UCI CFCCC)
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; HCC
Keywords: Hepatocellular Carcinoma; HCC; Cabozantinib; Ipilimumab; Nivolumab; TACE; transarterial chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Ipilimumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib with Ipilimumab/Nivolumab and TACE (Experimental): Subjects receive Cabozantinib 40 mg daily on days 1-28 of a 28 day cycle, this is to be started 7-14 days after the last TACE procedure.
  Nivolumab 480 mg IV on day 1 of a 28 day cycle (cycle 2 and beyond), this is to be started 7-14 days after the last TACE procedure.
  Nivolumab: 3mg/kg IV on day 1 of a 21 day cycle x 1 dose.
  Ipilimumab: 1 mg/kg on day 1 of a 21 day cycle x 1 dose
  TACE: Within 3-4 weeks of cycle 1 day 1; may be done up to 3 times (9-12 weeks total), the intervals between each TACE treatment can vary based on investigator's discretion
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Cabozantinib; Procedure: Transarterial Chemoembolization

INTERVENTIONS:
Drug: Nivolumab — Given IV
  Other Names: OPDIVO®
Drug: Ipilimumab — Given IV
  Other Names: YERVOY®
Drug: Cabozantinib — Given PO
  Other Names: CABOMETYX®; COMETRIQ
Procedure: Transarterial Chemoembolization — TACE treatment will be administered using either the DEB-TACE or cTACE modality in a series of up to 3 individual procedures within the 9-12 weeks following Day 21 (= cycle 1 day 21) of a patient's first infusion of nivolumab/ipilimumab. The first TACE treatment should start no more than 7 working days after being cycle 1 day 21.
  Other Names: TACE

SUMMARY:
This is a phase 2 single-arm, open-label clinical trial determining efficacy of cabozantinib in combination with ipilimumab/nivolumab and transarterial chemoembolization (TACE) in subjects with hepatocellular carcinoma (HCC). These are subjects who are not candidates for curative intent treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or radiographic diagnosis of hepatocellular carcinoma
* At least one lesion amenable to TACE treatment
* Child-Pugh A-B7 (B7 based on Albumin allowed)
* Not a candidate for resection or transplantation
* Age ≥ 18 years.
* Performance status: ECOG performance status ≤2
* Must have at least one measurable lesion (either untreated or progressed after previous locoregional treatment)
* Adequate organ and marrow function as defined below:

  1. Leukocytes ≥ 2,000/mcL
  2. absolute neutrophil count ≥ 1000/mcL
  3. platelets ≥ 60,000/mcl
  4. total bilirubin within normal institutional limits
  5. AST(SGOT)/ALT(SPGT) ≤ 3 X institutional upper limit of normal or ≤ 5 X if liver metastases are present
  6. creatinine <1.5ULN
  7. hemoglobin ≥ 8 g/dL
  8. Serum albumin ≥ 2.8 g/dL
  9. Urine protein/creatinine ration (UPCR) ≤ 1 mg/mg
* The effects of cabozantinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Based on its mechanism of action, ipilimumab can cause fetal harm when administered to a pregnant woman. Females of reproductive potential must use effective contraception during treatment with ipilimumab and for 3 months following the last dose of ipilimumab.

Based on its mechanism of action, nivolumab can cause fetal harm when administered to a pregnant woman. Females of reproductive potential must use effective contraception during treatment with nivolumab and for 5 months following the last dose of nivolumab.

1. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

1. Has not undergone a hysterectomy or bilateral oophorectomy; or
2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

   * Life expectancy of greater than 3 months
   * Ability to swallow tablets
   * Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Any type of previous systemic anti-cancer treatment
* All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to grade 1 or baseline
* Any locoregional treatment for HCC within 3 months
* Vp4 or Vp3 portal vein thrombus
* Extrahepatic disease
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, cabozantinib or other agents used in study.
* Concomitant anticoagulation with coumarin agents (eg, warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitors (e.g., rivaroxaban), or platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

  1. Prophylactic use of low-dose aspirin for cardioprotection (per local applicable guidelines) and low dose low molecular weight heparins (LMWH).
  2. Therapeutic doses of LMWH in subjects with a screening platelet count > 100,000/μL, without known brain metastases, and who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 28 days before the first dose of study treatment.
* Uncontrolled intercurrent illness including, but not limited to, the following conditions:

  1. ongoing or active infection
  2. symptomatic congestive heart failure
  3. uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment
  4. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before first dose
  5. unstable angina pectoris
  6. cardiac arrhythmia
  7. evidence of tumor invading GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
  8. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

     Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.
  9. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
  10. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  11. Lesions invading any major blood vessels. Subjects with lesions invading the intrahepatic vasculature, including portal vein, hepatic vein, and hepatic artery, are eligible.
  12. Other clinically significant disorders that would preclude safe study participation:

      1. Serious non-healing wound/ulcer/bone fracture
      2. Uncompensated/symptomatic hypothyroidism
      3. Moderate to severe hepatic impairment (Child-Pugh B or C)
  13. psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Prior treatment with cabozantinib
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.

Corrected QT (QTc) = QT / ∛RR

QT: duration of QT interval RR: duration of RR interval

Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early-stage prostate cancer, or curatively treated cervical carcinoma in-situ and not treated with systemic therapy.
* Inability to comply with study and follow-up procedures as judged by the Investigator
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants
* Has fibrolamellar HCC
* Has received prior cytotoxic, biologic or other systemic anticancer therapy including investigational agents within 4 weeks prior to randomization.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Has received a live vaccine within 30 days prior to the first dose of study intervention. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
* Has severe hypersensitivity (Grade ≥ 3) to nivolumab or cabozantinib and/or any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Has a history or current evidence of any condition (eg, known deficiency of the enzyme dihydropyrimidine dehydrogenase), therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Progression-free Survival at 6 Months | 6 months
  This is defined as the percentage of subjects who are free of progression 6 months after study treatment start. Progression is defined death, radiographic progression or clinical deterioration attributed disease progression as judged by an investigator. Radiographic progression is defined using the modified Response Evaluation Criteria in Solid Tumors Criteria (mRECIST), as a 20% increase in the sum of diameters of of viable (enhancing) target lesions and/or appearance of one or new lesions and/or unequivocal progression of existing non-target lesions.
Complete Response Rate | From date of registration until first date of disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  Complete Response (CR) is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.

SECONDARY OUTCOMES:
Overall Survival of Patients who Received Cabozantinib with Ipilimumab/Nivolumab and TACE | From date of registration for up to 18 months after last patient is enrolled or until death from any cause, whichever came first.
  To evaluate overall survival in patients with advanced gastric and gastroesophageal adenocarcinoma treated with this combination of cabozantinib and irinotecan.
Percentage of Grade 3-5 Adverse Events | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  To evaluate the tolerability of administering cabozantinib in combination with cabozantinib/nivolumab and TACE in patients with hepatocellular carcinoma from the start of treatment, duration of treatment and up to 4 weeks after completion of study treatment. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Progression Free Survival | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Conversion Rate to Resectable | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  Rate of subjects suitable for liver transplant according to the Milan criteria. Milan criteria is defined as single tumors ≤5 cm in diameter or no more than three tumors ≤3 cm in diameter single tumors ≤5 cm in diameter or no more than three tumors ≤3 cm in diameter

CONTACTS AND LOCATIONS:
Overall Officials: Farshid Dayyani, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States